CLINICAL TRIAL: NCT00672373
Title: A Double-Blind, Randomised, Parallel-Group Comparison of Extract of Ginkgo Biloba(EGB-761) Versus Placebo as Add-on Medication in Patients With Established Tardive Dyskinesia
Brief Title: Extract of Ginkgo Biloba and Tardive Dyskinesia
Acronym: EGBTD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing HuiLongGuan Hospital (Other)
Collaborators: Peking University (Other)
Responsible Party: Yun Long Tan, Beijing Hui-Long-Guan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EGB-ZWF-01; BJHLG-20061B0501900035
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2008-05-06 (Estimated); Status verified 2008-05

CONDITIONS: Tardive Dyskinesia; Schizophrenia
Keywords: Tardive Dyskinesia; Schizophrenia; Extract of Gingko Biloba
MeSH Terms: conditions — Tardive Dyskinesia; Schizophrenia | interventions — Ginkgo biloba extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Active treatment with EGb-761 capsules (80mg each capsule), 3 capsules each day for 12 weeks
  Interventions: Drug: Extract of Ginkgo Biloba (EGb-761 capsules)
- B (Placebo Comparator): Matching placebo treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Extract of Ginkgo Biloba (EGb-761 capsules) — EGb-761 240mg/d, 1 capsule(80mg) tid,po,12 weeks; Each capsule contains 19.6mg flavonol glycosides and 4.8mg terpene lactones.
  Other Names: YiKangNing
  Arms: A
Drug: Placebo — Wheat flour placebo capsule,1 capsule tid, po,12 weeks
  Arms: B

SUMMARY:
The purpose of this study is to determine whether Extract of Ginkgo Biloba is effective in the treatment on Tardive dyskinesia

DETAILED DESCRIPTION:
Tardive dyskinesia(TD) is a common complication of conventional antipsychotic treatment in subjects with schizophrenia. There is no established treatment for TD patients.This disorder remains a significant clinical problem for both patients and physicians for the foreseeable future.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 60yrs
* Meeting Diagnostic and Statistical Manual of Mental Diseases, Fourth Edition(DSM-IV) criteria for schizophrenia or schizo-affective disorder
* Abnormal Involuntary Movement Scale (AIMS) score ≥2.
* Patients from whom informed, written consent is obtained.
* Patients who have been on a fixed dose of antipsychotic medication for at least 4 weeks prior to trial entry.

Exclusion Criteria:

* Significant neurological disorder other than TD
* Substance abuse
* Significant other medical illness
* Psychiatric disorder not stabilised
* Pregnancy or lactation
* Take antioxidants(such as Vitamin C)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 157 (Actual)
Dates: Start 2006-12; Primary Completion 2007-05 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Change in the scores of Abnormal Involuntary Movement Scale (AIMS) | Baseline, 6th and 12th week

SECONDARY OUTCOMES:
Change in PANSS | Baseline, 6th and 12th week
Change in Simpson-Angus Rating Scales for EPS | Baseline, 6th and 12th
Change in cognitive function | Baseline and 12th week
Change in Udvalg for Kliniske Undersøgelser (UKU) Side Effect Rating Scale | Baseline, 6th and 12th week

CONTACTS AND LOCATIONS:
Overall Officials: Yunlong Tan, Phd, Principal Investigator — Beijing HuiLongGuan Hospital; Dongfeng Zhou, Professor, Study Chair — Institute of mental health, Peking University
Locations (1):
- Beijing Hui-Long-Guan Hospital, Beijing, China

REFERENCES:
- [Derived] Zhang WF, Tan YL, Zhang XY, Chan RC, Wu HR, Zhou DF. Extract of Ginkgo biloba treatment for tardive dyskinesia in schizophrenia: a randomized, double-blind, placebo-controlled trial. J Clin Psychiatry. 2011 May;72(5):615-21. doi: 10.4088/JCP.09m05125yel. Epub 2010 Sep 21. PMID 20868638